CLINICAL TRIAL: NCT01465984
Title: Comparison of IV Paracetamol With Intravenous Morphine Sulfate in Treatment of Acute Pain Due to Limb Trauma
Brief Title: Efficacy of Intravenous (IV) Paracetamol for Treatment of Acute Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACET1390; TUMS Thesis 1389 (Other Grant/Funding Number: TUMS)
Record Dates: First submitted 2011-11-02; First posted 2011-11-07 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Acute Pain
Keywords: Paracetamol; Morphine sulfates; Acute pain
MeSH Terms: conditions — Acute Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV Paracetamol (Experimental)
  Interventions: Drug: Paracetamol
- IV Morphine Sulfate (Active Comparator)
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Paracetamol — paracetamol , 1 gram Iv infusion Morphine Sulfate0.1 Mg/Kg Iv

SUMMARY:
The purpose of this study is to determine whether Iv paracetamol is as effective as Iv Morphine sulfate on control of the acute pain in Patient with limb trauma.

DETAILED DESCRIPTION:
Limb trauma is a painful condition that requires urgent analgesic treatment . Intravenous Opioids and NSAIDs are used extensively to control pain; both of them are with side effects. Paracetamol is a safe and effective analgesic that is used by oral or rectal routs for pain control, and in therapeutic doses has less side effects than Morphine and NSAIDs, and approved as a safe and effective analgesic in emergency department.

recently Iv Paracetamol has become available in European countries and also in Iran.

efficacy and safety of IV Paracetamol has been studied in post operation conditions and asserted but in emergency setting it has been studied only in renal colic situation.

Therefore, the investigators want to study the efficacy of IV Paracetamol in limb trauma and compare it with Iv Morphine sulfate.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute limb trauma
* Age>=18 years
* Acute pain of score 3 or greater on visual analogue scale

Exclusion Criteria:

* Unstable hemodynamic (Systolic blood pressure under 90 mmHg)
* Known sensitivity to opioids or paracetamol
* Any other known contraindication to Morphine Sulfate or Iv Paracetamol (including severe allergy to these drugs, acute bronchial asthma, upper respiratory tract obstruction)
* Previous administration of analgesic during 6 hours ago
* Pregnant women
* previous inclusion to the study
* diagnosed heart failure
* renal failure
* pulmonary failure or hepatic failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in pain severity/score | after 30 minutes

SECONDARY OUTCOMES:
Need for rescue analgesia | After 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Jalili, MD, Study Director — TUMS
Locations (1):
- TUMS, Tehran, Tehran Province, Iran